CLINICAL TRIAL: NCT07161219
Title: Implementation of New Exercise Protocols in Cardiac Rehabilitation.
Acronym: REVACARD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Dayez Martin, Principal investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: à compléter
Record Dates: First submitted 2025-03-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Heart Diseases; Cardiac Disease; Inspiratory Muscle Training
Keywords: heart failure; inspiratory muscles training
MeSH Terms: conditions — Heart Diseases; Heart Failure

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- intervention group (Experimental)
  Interventions: Device: inspiratory muscle training

INTERVENTIONS:
Device: inspiratory muscle training — inspiratory muscle training for intervention group
  Arms: intervention group

SUMMARY:
* Primary Objective: To evaluate the effects of complementary exercise protocols in cardiac rehabilitation (CR), such as inspiratory muscle training (IMT), by assessing inspiratory muscle strength.
* Secondary Objectives: To assess functional capacity, quality of life (QoL), and pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

- Patient meeting the conditions of the permanent life support agreement following hospitalization for a cardiac condition such as: acute myocardial infarction; coronary surgery; therapeutic percutaneous endovascular intervention on the coronary arteries, under medical imaging guidance; therapeutic percutaneous endovascular intervention on the heart, under medical imaging guidance; surgery for congenital or acquired heart malformation; surgery for valvular lesion; heart transplantation; resistant angina (to be specified by detailed history, medical history, and technical examinations, justifying multidisciplinary care); cardiomyopathy with left ventricular dysfunction (to be specified by detailed history, medical history, and technical examinations, justifying multidisciplinary care).

* Patient aged between 18 and 80 years.
* Patient capable of giving informed consent.
* Patient registered for permanent life support at the CuSL.
* Patient capable of understanding instructions in French. - Patient with prior medical consent and clinically stable.

Exclusion Criteria:

* - Minor (<18 years old).
* Pregnant woman.
* Patient unable to provide informed consent.
* Patient with cognitive, neurological, or orthopedic limitations.
* Patient with mobility or musculoskeletal difficulties incompatible with physical activity.
* Clinical instability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | 1 year